CLINICAL TRIAL: NCT02381756
Title: Ultrasound Evaluation of the Left Ventricular Systolic Function in Intensive Care Unit.
Brief Title: Ultrasound and Left Ventricular Systolic Function
Acronym: EFESE
Status: Terminated | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 2014-A01641-46
Record Dates: First submitted 2015-03-05; First posted 2015-03-06 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Dysfunction, Left Ventricular
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ultrasound — Cardiac echocardiography to determin the left ventricular ejection fraction by the biplane modified Simpson rule and by the calculation of the Strain Longitudinal Global by 2-D speckle tracking strain echocardiography

SUMMARY:
The aim of this study is to evaluate, in an intensive care unit, the reproducibility between two non-cardiologists operators and a cardiologist expert in echocardiogram, of the Simpson method and of the calculation of GLS for the evaluation of the systolic function of the left ventricle in critically ill patients intubated and ventilated.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients intubated and ventilated

Exclusion Criteria:

* Arrhythmia or variability of heart rate
* Technical impossibility to perform the ultrasound exam
* Known pregnancy or lactation
* Non-affiliation to a social security scheme (beneficiary or assignee)
* Patient under legal protection
* Patient refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients intubated and ventilated
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Reproducibility of measurements of the ejection fraction of the left ventricle by two measurement methods and reproducibility of myocardial strain measurements between operators | Baseline

SECONDARY OUTCOMES:
Area under the ROC curve of the value of myocardial strain (GLS) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Benyounes, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, Île-de-France Region, France